CLINICAL TRIAL: NCT06900179
Title: The Effectiveness of Augmented Reality Facilitated Education in Promoting Care Management of Malignant Fungating Wounds Among Oncology Nurses
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24MMHIS089e
Record Dates: First submitted 2024-12-24; First posted 2025-03-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-02

CONDITIONS: Nursing Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Reality (Experimental): Participants in the experimental group will receive an introduction to updated malignant fungating wound (MFWs) care guidelines and clinical applications, covering essential topics such as evidence-based wound management techniques, odor control, exudate handling, bleeding prevention, and pain management. Training will also address the identification and management of common MFWs-related complications, including infection. Additionally, participants will utilize the "MFWs with AR" program, engaging in simulated scenarios to enhance clinical reasoning and decision-making skills.
  Interventions: Other: MFWs with AR
- Classroom Teaching (Placebo Comparator): Classroom Teaching and Case Sharing Introduction to Updated MFWs Care Guidelines and Clinical Applications MFWs Wound Care Management of Common MFWs-Related Complications
  Interventions: Other: Classroom Teaching

INTERVENTIONS:
Other: MFWs with AR — MFWs with AR This study utilized MyWeb AR as the primary development platform to create an AR-enhanced teaching curriculum for malignant fungating wound (MFW) care. Based on the 2022 Clinical Care Guidelines for Malignant Fungating Wounds and expert input from oncology specialists, the content covers key aspects of MFW care, including wound assessment, symptom identification, and care principles such as odor control, exudate management, and infection prevention. The program uses 3D object elements and animations to create interactive AR scenarios, allowing participants to engage in simulated clinical decision-making and care management, thereby enhancing their skills in a safe and controlled environment.
  Arms: Augmented Reality
Other: Classroom Teaching — Classroom Teaching and Case Sharing Introduction to Updated MFWs Care Guidelines and Clinical Applications MFWs Wound Care Management of Common MFWs-Related Complications Case Sharing on MFWs Complication Management: Researchers
  Arms: Classroom Teaching

SUMMARY:
Malignant fungating wounds (MFWs) affect 5-14% of patients with advanced cancer, making them a common complication in this population. Characterized by symptoms such as foul odor, heavy exudate, bleeding, moderate to severe pain, and infection, MFWs cause significant physical discomfort and pose life-threatening risks while also leading to profound psychosocial issues, including shame and social isolation. These factors severely impact patients' quality of life, with half of those diagnosed surviving only six months on average.

However, clinical nursing staff often lack adequate knowledge and skills in managing MFWs, with an average accuracy rate of just 56.5%. Notable deficiencies exist in areas such as wound disinfection, odor control, and wound assessment, directly affecting the quality of patient care and highlighting an urgent need for specialized MFW training. Traditional MFW education often lacks real-life clinical scenarios and hands-on practice, resulting in a gap between learning and application and leaving learners ill-prepared for the complexities of clinical settings.

In contrast, augmented reality (AR) technology presents new possibilities for nursing education. AR can create highly simulated clinical environments where learners can safely practice complex clinical skills, enhancing clinical decision-making abilities. The implementation of AR-based training programs provides nursing staff with a more realistic and effective learning experience, allowing them to better address the challenges posed by MFWs and ultimately contributing to improvements in patient care and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Full-time nursing staff working in oncology wards at a teaching hospital in northern Taiwan
* Individuals willing to participate in the study and who have signed the informed consent form

Exclusion Criteria:

* Nursing staff not assigned to oncology-related wards
* Individuals expected to be unable to complete full participation in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
MFWs care Knowledge scale | 6months
  1. **MFWs Care Knowledge Scale** This study will assess MFWs care knowledge using the **MFWs Care Knowledge Scale**.
  The scale ranges from **0 to 100**, with higher scores indicating **better** knowledge levels.
  The assessment will be conducted at **baseline and post-intervention** to measure changes in MFWs care knowledge over time.

SECONDARY OUTCOMES:
Clinical Reasoning Scale | 6months
  This study will assess clinical reasoning ability using the Clinical Reasoning Scale. The scale ranges from 16 to 80, with higher scores representing better clinical reasoning ability. Measurements will be taken before and after the intervention to assess changes in clinical reasoning performance.

CONTACTS AND LOCATIONS:
Locations (1):
- MacKay Memorial Hosital, New Taipei City, New Taipei City, Taiwan